CLINICAL TRIAL: NCT04854551
Title: Opioid Modulation and Neural Reward Activation in Healthy Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 21-2886
Record Dates: First submitted 2021-04-08; First posted 2021-04-22 (Actual); Results first posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Alcohol Drinking; Opioid Use, Unspecified
MeSH Terms: conditions — Alcohol Drinking | interventions — Naltrexone

STUDY DESIGN:
Intervention Model Description: Participants will be counterbalanced for the order they undergo placebo and medication.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: capsule, double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo, Then Naltrexone (Experimental): Participants first received placebo capsules each day in a blister pack for 5 days. After a washout period of at least 3 days, they then received naltrexone capsules (matching placebo capsules) at 25mg/day for days 1 and 2 and then 50mg/day for days 3-5 for 5 days.
  Interventions: Drug: Naltrexone; Other: Placebo
- Naltrexone, Then Placebo (Experimental): Participants first received naltrexone capsules each day in a blister pack for 5 days. Days 1 and 2 were at 25mg/day, and days 3-5 were at 50mg/day. After a washout period of at least 3 days, they then received placebo capsules (matching naltrexone capsules) for 5 days.
  Interventions: Drug: Naltrexone; Other: Placebo

INTERVENTIONS:
Drug: Naltrexone — Naltrexone is an opioid antagonist with primary action at the mu opioid receptor.
Other: Placebo — Placebo will be used to control for expectancy effects

SUMMARY:
This is a double blind study of the effects of opioid antagonism on the brain's reward response. The investigators will recruit participants to undergo two scans, one on active medication and one on placebo. During the scan, the investigators will assess reward.

DETAILED DESCRIPTION:
The study will employ a crossover design. The study will use the monetary incentive delay task during functional MRI to assess reward. This task presents participants with cues indicating whether they are playing to win $5, win $0, or to avoid losing $5. This task has been well-validated to elicit activation in a key reward response area of the brain called the ventral striatum.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 35 years of age,
* Is a moderate drinker (i.e. consumes 1-14 drinks/week for males, or 1-7 drinks/week for females).

Exclusion Criteria:

* Non-drinker
* Positive result on urine drug screen or breathalyzer at the start of any study visit
* Inability to complete MRI (e.g. presence of ferromagnetic objects in body)
* Current use of medications that alter the hemodynamic response such as insulin
* History of trauma resulting in loss of consciousness longer than 15 minutes
* Currently taking opioid medications
* Pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Gowin, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators would either upload to an online repository or share directly with individuals wishing to access it.

REFERENCES:
- [Derived] Gowin JL, Sloan ME, Kirk-Provencher KT, Rosenblatt SL, Penner AE, Stangl BL, Byrd ND, Swan JE, Ramchandani VA. Opioid receptor antagonism and neural response to monetary rewards: Pilot studies in light and heavy alcohol users. J Psychopharmacol. 2023 Sep;37(9):937-941. doi: 10.1177/02698811231191707. Epub 2023 Aug 2. PMID 37530456

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Adults: Placebo First, Then Naltrexone: This arm will receive placebo first, then active medication second
  Naltrexone: Naltrexone is an opioid antagonist with primary action at the mu opioid receptor.
  Placebo: Placebo will be used to control for expectancy effects
- Healthy Adults: Active Medication First, Then Placebo: This arm will receive active medication first, then placebo second
  Naltrexone: Naltrexone is an opioid antagonist with primary action at the mu opioid receptor.
  Placebo: Placebo will be used to control for expectancy effects
Period: Overall Study
Arm/Group | Healthy Adults: Placebo First, Then Naltrexone | Healthy Adults: Active Medication First, Then Placebo
Started | 7 | 6
Completed | 6 | 5
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Healthy young adults
Groups:
- Healthy Adults: Placebo First: This arm will receive placebo first, then active medication second
  Naltrexone: Naltrexone is an opioid antagonist with primary action at the mu opioid receptor.
  Placebo: Placebo will be used to control for expectancy effects
- Healthy Adults: Active Medication First: This arm will receive active medication first, then placebo second
  Naltrexone: Naltrexone is an opioid antagonist with primary action at the mu opioid receptor.
  Placebo: Placebo will be used to control for expectancy effects
- Total: Total of all reporting groups
Arm/Group | Healthy Adults: Placebo First | Healthy Adults: Active Medication First | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.8 (4.4) | 24.0 (4.4) | 24.2 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Brain Activation to Reward Between Placebo and Active Medication
Description: Percent signal change relative to baseline in the nucleus accumbens during cue to win $5 as assessed during functional MRI. Higher values of percent signal change indicate greater activation to reward. We will compare the active medication condition to the placebo, establishing whether there is a difference between the conditions.
Time Frame: one week
Population: The participants who completed the study were analyzed. They were all healthy adults who met inclusion/exclusion criteria.
Measure: Mean (Standard Deviation); unit: percentage signal change
Groups:
- Naltrexone: Participants who received Naltrexone capsules for 5 days (25mg for days 1 and 2, then 50mg for days 3, 4, and 5) before either the first or second scanning session.
- Placebo: Participants who received Placebo capsules for 5 days before either the first or second scanning session
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 11 | 11
percentage signal change | 0.25 (0.09) | 0.26 (0.10)

2. Secondary Outcome: Alcohol Value
Description: Maximum alcohol expenditure, or Omax, is the maximum amount of money that a person will pay for alcohol in a hypothetical alcohol consumption task called the "Alcohol Purchase Task". Higher values of Omax indicate that a person values consuming alcohol at a greater level.
Time Frame: one week
Population: Healthy adults who completed the study
Measure: Mean (Standard Deviation); unit: Dollars
Groups:
- Placebo: Participants who received Placebo capsules before either the first or second scanning session.
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 11 | 11
Dollars | 19.4 (14.8) | 19.9 (17.4)

3. Secondary Outcome: Brain Activation to Emotion Regulation
Description: Percent signal change from baseline in the amygdala during trials to regulate emotion relative to trials to passively experience emotion during a functional MRI scan. Cues will be negative images, and instructions will be either "decrease" or "look".
Time Frame: one week
Measure: Mean (Standard Deviation); unit: percentage signal change
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 11 | 11
percentage signal change | 0.1 (0.1) | 0.1 (0.1)

ADVERSE EVENTS:
Time Frame: 1 week
Description: Self report
Arm/Group | Naltrexone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT04854551/Prot_SAP_000.pdf